CLINICAL TRIAL: NCT06344468
Title: The Effect of Early Mobilization on Sleep, Physiological Parameters, and Length of Stay in ICU: A Randomized Controlled Study
Brief Title: The Effect of Early Mobilization on Sleep, Physiological Parameters, and Length of Stay in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ahmet Sen, Registered Nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 531393
Record Dates: First submitted 2024-03-07; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Early Mobilization; Sleep Quality; Critical Care; Nursing Caries
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Early mobilization began after discontinuation of sedation and resolution of its effects within the first 12 hours. During early mobilization, physiological parameters (respiratory rate, SpO2, heart rate, blood pressure, body temperature, pain) were evaluated and recorded in the supine and semi-fowler positions for in-bed mobilization assessment. For out-of-bed mobilization, physiological parameters were determined and recorded while the patient was in a sitting position, with the head elevated at 45° before mobilization.
  With the assistance of a nurse, the patient was guided to sit on the edge of the bed, stand up with support, sit on a chair next to the bed, and record respiratory rate, SpO2, heart rate, blood pressure, body temperature, and pain levels at 1, 5, and 10 minutes while sitting on the chair. Similar procedures were repeated during patient mobilization at 24 and 36 hours.
  Interventions: Other: Early Mobilization
- Control Group (No Intervention): They underwent routine/standard postoperative mobilization procedures. Accordingly, patients were mobilized within the first 24 hours post-surgery, and during in-bed mobilization, physiological parameters (respiratory rate, SpO2, heart rate, blood pressure, body temperature, pain) were evaluated in the supine and semi-fowler positions.During out-of-bed mobilization, physiological parameters (respiratory rate, SpO2, heart rate, blood pressure, body temperature, pain) were determined.
  Respiratory parameters were frequently evaluated at intervals of up to 4 hours using arterial blood gas analysis. The patient was assisted by a nurse to sit on the edge of the bed, stand up with support, sit on a chair next to the bed, and record respiratory rate, SpO2, heart rate, blood pressure, body temperature, and pain levels at 1, 5, and 10 minutes while sitting on the chair. These data were then evaluated internally. Similar procedures were repeated during patient mobilization at 24 and 36 hours.

INTERVENTIONS:
Other: Early Mobilization — Essentially, early mobilization practices consist of two parts: in-bed and out-of-bed. In-bed mobilization; Active-passive joint range of motion (ROM) Exercises include raising the head in bed, turning in bed, in-bed exercises and sitting at the end of the bed. Out-of-bed mobilization includes the process of transferring from bed to chair, standing up, and returning to bed after standing up. In studies conducted on cardiac surgery, the early mobilization period is the first 12 hours.
  Arms: Experimental Group

SUMMARY:
The goal of this is randomized controlled study to examine the effect of early mobilization on sleep, physiological parameters, and length of stay in the intensive care unit (ICU).

The hypothesis are:

Hypothesis I: Early mobilization positively affects the sleep quality of patients.

Hypothesis II: Early mobilization positively affects the physiological parameters of patients (respiratory rate, heart rate, blood pressure, body temperature, pain).

Hypothesis III: Early mobilization shortens the length of stay of patients in the intensive care unit (ICU).

Early mobilization will begin in the experimental group after sedation is discontinued within the first 12 hours and its effects disappear. In early mobilization, in the evaluation of in-bed mobilization, physiological parameters (respiratory rate, sPO 2, heart rate, blood pressure, body temperature, pain) will be evaluated and recorded in the supine, semi-fowler position. In out-of-bed mobilization, the patient's physiological parameters (respiratory rate, sPO 2, heart rate, blood pressure, body temperature, pain) will be determined and recorded before mobilization and when the head is in a 45˚ upward position. Surgical wounds and dressing areas, if any, are protected, drains are identified, care is taken not to remove equipment such as urinary catheters or nasogastric tubes, when the patient is seated on the edge of the bed with the help of a nurse, when he/she is stood up next to the bed with the support of the nurse, when he/she is made to sit in a chair next to the bed and when he/she is in a chair. While sitting, 1st minute, 5th minute, 10th minute respiratory rate, sPO2, heart rate, blood pressure, body temperature values and pain levels will be recorded and these data will be evaluated on their own. During mobilization, if the patient develops chest pain, arrhythmia, hypertension (systolic pressure>160 mmHg), or hypotension (systolic pressure<90 mmHg), tachypnea, or hypoxia, a break will be taken and the physician will be consulted. The same procedures will be repeated during the mobilization of the patient in the first 24-36 hours and the necessary records will be made by the researcher.

Control Group:

After admission to the Cardiovascular Surgery ICU, the type, purpose and implementation process of the study will be explained to the patients, and a routine/standard postoperative mobilization procedure will be applied to the patients in the control group. Accordingly, patients will be mobilized in the first 24 hours after surgery, and in the evaluation of in-bed mobilization, their physiological parameters (respiratory rate, sPO 2, heart rate, blood pressure, body temperature, pain) will be evaluated and recorded in the supine, semi-fowler position. In out-of-bed mobilization, the patient's physiological parameters (respiratory rate, sPO 2, heart rate, blood pressure, body temperature, pain) will be determined and recorded before mobilization and when the head is in a 45˚ upward position. Again, arterial blood gas monitoring of the patients in the control group will be performed at maximum 4-hour intervals, and respiratory parameters will be frequently evaluated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older,
* Have been in the ICU for at least 36 hours,
* Be independent in their mobility activities,
* Maintain respiratory activity without being dependent on a device/equipment,
* Have a Glasgow Coma Scale score of at least 15,
* Have sedation discontinued within the first 6 hours.

Exclusion Criteria:

* Be fully sedated,
* Have neurological or orthopedic conditions that could create contraindications (such as cerebrovascular events, circulatory disorders, pulmonary embolism),
* Be unable to tolerate mobilization (severe bradycardia, arrhythmia, chest pain, hypotension, hypertension, tachypnea, SaO2 <90%, etc.),
* Have a Glasgow Coma Scale score below 15,
* Be dependent on mobility activities before surgery,
* Use sleep medication and experience sleep problems before surgery,
* Have extubation not performed within the first 24 hours after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
The length of stay of patients in the intensive care unit | At least 2 days, up to 12 months.
  The length of stay of a patient in the intensive care unit refers to the duration from the patient's admission to the intensive care unit until their discharge

SECONDARY OUTCOMES:
The Richards-Campbell Sleep Questionnaire (RCSQ) | At the moment the patient is admitted to the hospital, at the 12th hour in the Intensive Care Unit (ICU), at the 24th hour in the ICU and at the 36th hour in the ICU.
  The Richards Campbell Sleep Scale, developed by Kathy C. Richards in 1987, aims to determine patients' nighttime sleep depth, sleep onset latency, wakefulness during the night, time awake after sleep onset, and overall sleep quality. The scale consists of 6 items, with participants asked to rate each item on a scale from 0 to 100. Scores ranging from 0 to 25 indicate very poor sleep, while scores between 75 and 100 indicate very good sleep. As the total score on the scale increases, sleep quality also improves.
The Glasgow Coma Scale (GCS) | At the moment the patient is admitted to the hospital, at the 12th hour in the Intensive Care Unit (ICU), at the 24th hour in the ICU, and at the 36th hour in the ICU.
  The Glasgow Coma Scale (GCS) was developed by Teasdale and Jennett in 1974. GCS is one of the assessment tools used to define, classify, and eliminate the risk of incomplete or incorrect evaluation of levels of consciousness. With GCS, patients' eye opening, verbal, and motor responses are assessed. The total score on the scale is 15, with 15 points indicating full alertness and awareness. The lowest score on the scale is 3, indicating deep coma. According to GCS, a score of 8 or below indicates that the patient is unconscious and in a coma, requiring intensive care.
Physiological Parameter - for the experimental group | At the moment of extubation, during the first mobilization within the first 12 hours after surgery, 15, 30, and 60 minutes after mobilization, and at the 12th and 24th hours in intensive care.
  Researchers have developed a physiological parameter monitoring form to track and record patients' physiological parameters before and after surgery. The form includes minute respiratory rate, sPO2, PaO2, PaCO2, heart rate, blood pressure, body temperature, and pain values. The patient's minute respiratory rate, sPO2, heart rate, blood pressure, and body temperature will be monitored using monitoring devices. PaO2 and PaCO2 values will be monitored during the patient's intensive care process using arterial blood gas analysis. The patient's pain intensity will be evaluated using a Visual Analog Scale (VAS) ranging from 0 for no pain to 10 for severe pain.
Physiological Parameter - for the control group | At the moment of extubation, during the first mobilization within the first 12-24 hours after surgery, 15, 30, and 60 minutes after mobilization, and at the 12th and 24th hours in intensive care
  Researchers have developed a physiological parameter monitoring form to track and record patients' physiological parameters before and after surgery. The form includes minute respiratory rate, sPO2, PaO2, PaCO2, heart rate, blood pressure, body temperature, and pain values. The patient's minute respiratory rate, sPO2, heart rate, blood pressure, and body temperature will be monitored using monitoring devices. PaO2 and PaCO2 values will be monitored during the patient's intensive care process using arterial blood gas analysis. The patient's pain intensity will be evaluated using a Visual Analog Scale (VAS) ranging from 0 for no pain to 10 for severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University-Cerrahpaşa Cerrahpaşa School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ashkenazy S, DeKeyser-Ganz F. Assessment of the reliability and validity of the Comfort Scale for adult intensive care patients. Heart Lung. 2011 May-Jun;40(3):e44-51. doi: 10.1016/j.hrtlng.2009.12.011. Epub 2010 Apr 8. PMID 20561865
- [Result] Taito S, Shime N, Ota K, Yasuda H. Early mobilization of mechanically ventilated patients in the intensive care unit. J Intensive Care. 2016 Jul 29;4:50. doi: 10.1186/s40560-016-0179-7. eCollection 2016. PMID 27478617
- [Result] Chen B, You X, Lin Y, Dong D, Xie X, Zheng X, Li D, Lin W. A systematic review and meta-analysis of the effects of early mobilization therapy in patients after cardiac surgery: A protocol for systematic review. Medicine (Baltimore). 2020 Jan;99(4):e18843. doi: 10.1097/MD.0000000000018843. PMID 31977881
- [Result] TEAM Study Investigators and the ANZICS Clinical Trials Group; Hodgson CL, Bailey M, Bellomo R, Brickell K, Broadley T, Buhr H, Gabbe BJ, Gould DW, Harrold M, Higgins AM, Hurford S, Iwashyna TJ, Serpa Neto A, Nichol AD, Presneill JJ, Schaller SJ, Sivasuthan J, Tipping CJ, Webb S, Young PJ. Early Active Mobilization during Mechanical Ventilation in the ICU. N Engl J Med. 2022 Nov 10;387(19):1747-1758. doi: 10.1056/NEJMoa2209083. Epub 2022 Oct 26. PMID 36286256
- [Result] Menges D, Seiler B, Tomonaga Y, Schwenkglenks M, Puhan MA, Yebyo HG. Systematic early versus late mobilization or standard early mobilization in mechanically ventilated adult ICU patients: systematic review and meta-analysis. Crit Care. 2021 Jan 6;25(1):16. doi: 10.1186/s13054-020-03446-9. PMID 33407707
- [Result] Norimoto M, Yamashita M, Yamaoka A, Yamashita K, Abe K, Eguchi Y, Furuya T, Orita S, Inage K, Shiga Y, Maki S, Umimura T, Sato T, Sato M, Enomoto K, Takaoka H, Hozumi T, Mizuki N, Kim G, Ohtori S. Early mobilization reduces the medical care cost and the risk of disuse syndrome in patients with acute osteoporotic vertebral fractures. J Clin Neurosci. 2021 Nov;93:155-159. doi: 10.1016/j.jocn.2021.09.011. Epub 2021 Sep 20. PMID 34656240
- [Result] Rezvani H, Esmaeili M, Maroufizadeh S, Rahimi B. The Effect of Early Mobilization on Respiratory Parameters of Mechanically Ventilated Patients With Respiratory Failure. Crit Care Nurs Q. 2022 Jan-Mar 01;45(1):74-82. doi: 10.1097/CNQ.0000000000000390. PMID 34818300
- See also: Related Info — https://doi.org/10.12681/healthresj.28161